CLINICAL TRIAL: NCT01101789
Title: Triclosan Coated Suture Wound Closure for Peripheral Vascular Surgery: a Prospective Multicenter Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Karelia Central Hospital (Other)
Responsible Party: Principal Investigator, Sanna Kouhia, MD, North Karelia Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NKCH-surg-006
Record Dates: First submitted 2010-04-08; First posted 2010-04-12 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Surgical Wound Infection
Keywords: surgical wound infection; triclosan-coated suture
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- triclosan (Active Comparator): triclosan-coated sutures
  Interventions: Procedure: triclosan coated suture for surgical wound closure
- control (Placebo Comparator): sutures without triclosan-coating
  Interventions: Procedure: regular sutures for surgical wound closure

INTERVENTIONS:
Procedure: triclosan coated suture for surgical wound closure — triclosan coated suture for surgical wound closure
  Arms: triclosan
Procedure: regular sutures for surgical wound closure
  Arms: control

SUMMARY:
This is a prospective randomized multicenter study which purpose is to determine whether triclosan-coated sutures for wound closure after lower limb vascular surgery would reduce the incidence of surgical wound infections.

ELIGIBILITY:
Inclusion Criteria:

* patient undergoing peripheral vascular surgery procedure

Exclusion Criteria:

* patients refusal

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2010-04; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
surgical wound infection | one month after surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Turtiainen, MD, Study Director — North Karelia Central Hospital; Kimmo Makinen, Principal Investigator — Kuopio University Hospital; Maarit Venermo, Principal Investigator — Helsinki University Central Hospital; Eija Saimanen, Principal Investigator — South Carelia Central Hospital; Ilkka Uurto, Study Director — Tampere University Hospital
Locations (1):
- North Carelia central hospital, Joensuu, Joensuu, Finland